CLINICAL TRIAL: NCT01481168
Title: Adenosine Testing to DEtermine the Need for Pacing Therapy With the Additional Use of an Implantable Loop Recorder (ADEPT-ILR Study). The Efficacy of Permanent Pacing in Patients With Syncope and a Positive Intravenous Adenosine Test: a Randomised, Double-blind, Placebo-controlled, Cross-over Trial.
Brief Title: Adenosine Testing to DEtermine the Need for Pacing Therapy
Acronym: ADEPT-ILR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Newcastle-upon-Tyne Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 5883; FS/11/13/28690 (Other Grant/Funding Number: British Heart Foundation)
Record Dates: First submitted 2011-11-22; First posted 2011-11-29 (Estimated); Last update posted 2017-11-20 (Actual); Status verified 2017-11

CONDITIONS: Syncope
MeSH Terms: conditions — Syncope

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Pacemaker "on" (Active Comparator): DDD+/-R pacing
  Interventions: Device: Pacemaker implantation (Medtronic)
- Pacemaker "off" (Placebo Comparator): ODO pacing
  Interventions: Device: Pacemaker implantation (Medtronic)
- Implantable Loop Recorder (Experimental): Implantable loop recorder in adenosine test negative patients
  Interventions: Device: Implantable Loop Recorder (Medtronic)

INTERVENTIONS:
Device: Pacemaker implantation (Medtronic) — DDD+/-R pacing
  Other Names: Medtronic DDD+/-R pacemakers
  Arms: Pacemaker "on"
Device: Pacemaker implantation (Medtronic) — ODO pacing
  Other Names: Medtronic DDR+/-R pacemakers.
  Arms: Pacemaker "off"
Device: Implantable Loop Recorder (Medtronic) — Loop recorder implantation
  Other Names: Medtronic Reveal DX or XT
  Arms: Implantable Loop Recorder

SUMMARY:
The purpose of this study is to determine whether or not the intravenous adenosine test readily identifies patients with unexplained syncope who would benefit from permanent pacemaker implantation.

DETAILED DESCRIPTION:
The investigation of syncope (transient loss of consciousness with loss of postural tone, collapse and spontaneous recovery) varies widely, is often lengthy and frequently expensive. The intravenous adenosine test has been used in the investigation of syncope and is cheap, safe and free of serious side effects. However, it is unclear what diagnosis the test unearths. There is some evidence that the test readily identifies bradycardia pacing indications.

In this study we plan to perform the adenosine test and implant a pacemaker should the test be positive. In half of the patients we will turn the pacemaker "on" and in the other half the pacemaker "off". The groups will swap over after six months. During this time we will assess the number of syncopal episodes. Also, in those who have a negative adenosine test we will implant a loop recorder to try to discover the cause of syncope.

ELIGIBILITY:
Inclusion Criteria:

* Episode of syncope
* Patient has provided written informed consent for participation in the study prior to any study specific procedures
* Male or female
* Age > 40 years
* No cause of syncope clearly identified on clinical examination, lying and standing blood pressure measurements and standard 12 lead ECG.

Exclusion Criteria:

* Asthma or chronic obstructive pulmonary disease
* Severe coronary disease (myocardial infarction within 3 months, known coronary stenosis >70%, NYHA heart failure or angina symptoms Class III or IV)
* Known severe cerebrovascular disease or known significant internal carotid artery stenosis (>70%)
* Prolonged corrected QT interval
* Unablated accessory pathway
* Pregnancy or lactation
* Use of dipyridamole or any rate-limiting medication that cannot be safely discontinued
* Hypertrophic cardiomyopathy
* Cardiac transplantation
* Concurrent participation in another investigational study or trial
* Inability to give informed consent; carer/proxy assent will be allowed in this study
* Cause of syncope established from initial clinical history and examination, lying and standing blood pressure and ECG

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2012-04-12 (Actual); Primary Completion 2017-01-26 (Actual); Study Completion 2017-01-26 (Actual)

PRIMARY OUTCOMES:
Syncope Burden | 12 months
  Syncope Burden as measured by number of syncopal episodes and recorded by weekly postal patient diaries with telephone reminders to ensure adequate return

SECONDARY OUTCOMES:
Time to first syncope | 12 months
  Time to first syncope
Number of patients with recurrent syncope | 12 months
  Number of patients with >1 episodes of syncope
Quality of life | 12 months
  Quality of life as measured via the condition-specific instrument the Impact of Syncope on Quality of Life questionnaire with general health-related quality of life measured via the WHOQoL-Brief and WHOQoL-Old instruments
Health economic analysis | 12 months
  Costs and benefits of the intervention to health and social services. (i) Use of EQ-5D questionnaire to establish the cost per Quality Adjusted Life Year (QALY) (ii) The analysis will include the patients described above as well as a historical comparator group of consecutive patients derived from the database held by the Falls and Syncope Service who have not undergone adenosine testing. This group is particularly important to establish the utility of adenosine testing in the diagnosis of unexplained syncope.
ECG diagnosis on ILR following syncopal episode in adenosine negative group | 12 months
  ECG diagnosis on ILR following syncopal episode in intravenous adenosine test negative group

CONTACTS AND LOCATIONS:
Overall Officials: Steve W Parry, PhD, MBBS, MRCP, BSc, Principal Investigator — Institue of Ageing and Health, University of Newcastle; Chris J Pummer, PhD, MRCP, BMBCh, BSc, Principal Investigator — Newcastle upon Tyne Hospitals NHS FOundation Trust
Locations (2):
- United Kingdom (2):
  - Royal Victoria Infirmary, Newcastle upon Tyne, Tyne and Wear
  - Feeeman Hospital, Newcastle upon Tyne, Tyne and Wear